CLINICAL TRIAL: NCT03298906
Title: A Fixed-sequence, Open-label Study to Assess the Effect of Ticlopidine on the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Healthy Subjects
Brief Title: A Study to Assess the Effect of Ticlopidine on the Pharmacokinetics, Safety, and Tolerability of Intranasally Administered Esketamine in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CR108377; 54135419TRD1020 (Other: Janssen Research & Development, LLC); 2017-003174-14 (EudraCT Number)
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Healthy
MeSH Terms: interventions — Esketamine; Ticlopidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Esketamine + Ticlopidine (Experimental): Participants will self-administer one 14 milligram (mg) spray of intranasal esketamine into each nostril at Time 0 and again 5 minutes later on Day 1, a total dose of 56 mg (Treatment A) in Treatment Period 1. After that participants will receive 250 mg of ticlopidine tablets orally twice daily on Day -9 through Day 1, and will self-administer one 14 mg spray of intranasal esketamine into each nostril at Time 0 and again 5 minutes later in the morning of Day 1, a total dose of 56 mg (Treatment B) in Treatment Period 2. A washout period of greater than or equal to (>=)10 days will separate the esketamine self-administrations between 2 treatment periods.
  Interventions: Drug: Esketamine; Drug: Ticlopidine

INTERVENTIONS:
Drug: Esketamine — Participants will self-administer one intranasal spray of 14 mg esketamine at Time 0 and again 5 minutes later on Day 1, a total dose of 56 mg in Treatment Period 1 and 2.
  Other Names: JNJ-54135419
Drug: Ticlopidine — Participants will receive 250 mg ticlopidine tablets orally twice daily on Day -9 through Day 1 in Treatment Period 2.

SUMMARY:
The purpose of this study is to evaluate the effects of ticlopidine on the pharmacokinetics (PK) of intranasally administered esketamine.

ELIGIBILITY:
Inclusion Criteria:

* Be healthy on the basis of physical examination, medical history, vital signs, and 12-lead electrocardiogram (ECG) performed at screening
* A woman must be either:

  1. Not of childbearing potential defined as:

     1. postmenopausal (it is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone [FSH] level [greater than {>}40 International Unit per Liter {IU/L} or milliinternational Unit per milliliter {mIU/mL}] in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy, however in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient)
     2. permanently sterile (permanent sterilization methods include hysterectomy, bilateral salpingectomy, bilateral tubal occlusion/ligation procedures, and bilateral oophorectomy)
  2. Of childbearing potential, heterosexually active, and

     1. practicing a highly effective method of contraception (failure rate of less than [<]1 percent [%] per year when used consistently and correctly)
     2. agree to remain on a highly effective method throughout the study and for at least 6 weeks after the last dose of study drug
* For women, must have a negative serum Beta- human chorionic gonadotropin (Beta-hCG) pregnancy test at screening
* During the study and for a minimum of 1 spermatogenesis cycle (defined as approximately 90 days) after receiving the last dose of intranasal study medication, a man who is sexually active with a woman of childbearing potential

  1. must be practicing a highly effective method of contraception with his female partner
  2. must use a condom if his partner is pregnant, and
  3. must agree not to donate sperm
* Have a creatinine clearance greater than or equal to (>=) 60 milliliter per minute (mL/min) (calculated using the Cockcroft-Gault formula) at screening

Exclusion Criteria:

* Has a current significant psychiatric disorder including but not limited to psychotic, bipolar, major depressive, or anxiety disorder
* Has a clinically significant medical illness including (but not limited to) cardiac arrhythmias or other cardiac disease, hematologic disease, coagulation disorders (including any abnormal bleeding or blood dyscrasias), lipid abnormalities, significant pulmonary disease, including bronchospastic respiratory disease, diabetes mellitus, renal or hepatic insufficiency, thyroid disease, neurologic disease, infection, hypertension or vascular disorders, kidney or urinary tract disturbances, sleep apnea, myasthenia gravis, or any other illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results. Participants with medical conditions that are stable with treatment may be included and should be discussed with the medical monitor before inclusion
* Has clinically significant abnormal values for hematology, serum chemistry, or urinalysis at screening as deemed appropriate by the investigator
* Has any contraindication to the use of ticlopidine, ketamine, or esketamine per prescribing information
* Has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at screening

Ages: 18 Years to 58 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2017-09-26 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Esketamine | Day 1: 0 (pre-dose), 7, 12, 20, 30, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18, 24 and 30 hours post-dose
  The Cmax is the maximum observed plasma concentration.
Area Under the Plasma Concentration-time Curve From Time Zero to Infinite Time (AUC [0-infinity]) of Esketamine | Day 1: 0 (pre-dose), 7, 12, 20, 30, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18, 24 and 30 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(0-last) and C(0-last)/lambda(z), wherein AUC(0-last) is area under the plasma concentration time curve from time zero to last quantifiable time; C(0-last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-time Curve From Time Zero to time of Last Quantifiable Concentration (AUC [0-last]) of Esketamine | Day 1: 0 (pre-dose), 7, 12, 20, 30, 40, 50 minutes; 1, 1.25, 1.5, 2, 3, 4, 6, 9, 12, 18, 24 and 30 hours post-dose
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable concentration.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events (AEs) as a measure of Safety and Tolerability | From signing of the informed consent form (ICF) onwards until the participant's last study-related activity (Approximately up to 8 weeks)
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Clinical Pharmacology Unit, Merksem, Belgium